CLINICAL TRIAL: NCT07256925
Title: LEVEL-UP Turkish Adult Outpatient Screening Study
Brief Title: Malnutrition Screening Study
Status: Recruiting | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA34
Record Dates: First submitted 2025-11-21; First posted 2025-12-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Malnutrition, Calorie; Sarcopenia
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital Clinics: Oncology, Neurology and Geriatric

SUMMARY:
This is a non-interventional, cross-sectional, non-randomized, observational study to screen for the risk of malnutrition and sarcopenia in outpatients aged 18 and over who attend hospital clinics for any reason in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Participant has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and provided other applicable privacy regulation authorization (if applicable) prior to any participation in the study.
* Participant is ≥ 18 years of age who attend hospital clinics (medical and radiation oncology, neurology, and geriatrics clinics) as an outpatient for any reason.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants attending medical and radiation oncology, neurology, and geriatrics outpatient hospital clinics in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Malnutrition Risk | Screening Study Day 1
  Measured via R-MAPP Screening Questionnaire completed by participant interview.
Sarcopenia Risk | Screening Study Day 1
  Measured via R-MAPP Screening Questionnaire completed by participant interview.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Screening Study Day 1
  Calculated as weight (kg)/height (m)2
Calf Circumference | Screening Study Day 1
  Measured in cm
Hand Grip Strength | Screening Study Day 1
  Measured in kg by hand grip dynamometer
Biochemical Parameters | Screening Study Day 1
  Albumin, CRP and Vitamin D
Health Care Utilization | Screening Study Day 1
  Number of Outpatient and Hospitalization Admissions during the past 6 months.
Nutrition Treatment | Screening Study Day 1
  Number of participants referred for medical nutrition treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aysugul Alptekin, MD, Study Chair — Abbott Nutrition
Locations (1):
- Necmettin Erbakan University Faculty of Medicine General Surgery, Meram, Konya, Turkey (Türkiye)